CLINICAL TRIAL: NCT04869514
Title: Does Spinal Manipulation Therapy Impact Lumbar Proprioception? A Double-blind Randomized Controlled Trial Examining the Influence of Spinal Manipulative Therapy (SMT) Versus a Sham and Non-sham Control Intervention on Proprioceptive Function
Brief Title: Does Spinal Manipulation Therapy Impact Lumbar Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Michael Meier, Principal Investigator, Balgrist University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Project Nexus
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Manipulation, Psychologic; Proprioception; Vibration; Exposure
MeSH Terms: interventions — Manipulation, Spinal

STUDY DESIGN:
Intervention Model Description: The study design consists of a four-arm (1:1:1:1 ratio) randomized controlled trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The data collection and analysis will be conducted by a research assistant blind to treatment allocation. The study subjects will be blinded with respect to the hypothesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- either lumbar manipulation (LMANIP) (Active Comparator): LMANIP will consist of high velocity low amplitude (HVLA) SMT at the L4/L5 motion segment. LMANIP consists of two HVLA impulses, applied in side-posture on the right and left side (order pseudorandomized).
  Interventions: Procedure: spinal manipulation
- thoracic manipulation (TMANIP) (Active Comparator): TMANIP will consist of high velocity low amplitude (HVLA) SMT at the T4/5 motion segment. TMANIP consists of supine SMT to the right and left (order pseudorandomized) using a thenar contact at facet joint level T4/5
  Interventions: Procedure: spinal manipulation
- lumbar mobilisation (LMOB) (Sham Comparator): LMOB will be applied with the same positioning as in the LMANIP procedure, but instead of a thrust, a slow, a slow, passive mobilization without impulse will be applied
  Interventions: Procedure: spinal manipulation
- No intervention (No Intervention): A natural history arm will serve to further control for potential specific and non-specific effects of TMANIP and LMOB. Subject will rest in side-lying position for the same duration as during the active interventions.

INTERVENTIONS:
Procedure: spinal manipulation — intervention will consist of either lumbar manipulation, thoracic manipulation or lumbar mobilisation
  Arms: either lumbar manipulation (LMANIP); lumbar mobilisation (LMOB); thoracic manipulation (TMANIP)

SUMMARY:
Spinal manipulation therapy (SMT) has long been a component of manual therapy and physical rehabilitation programs, especially as a modality for pain relief. However, the underlying physiological mechanisms for manipulation-related pain relief and functional improvement remain largely unexplored. To promote targeted treatments for musculoskeletal conditions and to better identify the indication and scope of SMT, its mechanisms must be better understood.

DETAILED DESCRIPTION:
Manual therapy is widely used by patients with back pain with about 75% of patients consulting either a chiropractor, physiotherapist or osteopath. Often used manual therapies include spinal manipulative therapy (SMT), which is recommended in several clinical guidelines for management of back pain, mostly for acute low back pain (LBP) but also for chronic LBP. Despite the clinical benefits of SMT, the mechanisms underlying its effectiveness are poorly understood. Several mechanisms of action have been proposed including biomechanical and neurophysiological effects observed on spinal and supraspinal levels with unclear relationship to potential analgesic effects. Furthermore, non-specific effects such as placebo effects can strongly influence treatment outcomes and are difficult to control as consensus is lacking regarding the "active" agent of SMT, making it challenging to design an adequately controlled and blinded study.

A potential biological mechanism underlying the effectiveness of SMT might be related to sustained changes in lumbar proprioceptive function following repeated mechanical pressure on spinal tissues. In support of this, evidence from animal studies indicates that SMT comparable forces applied to the spine increase the discharge frequency of proprioceptive afferents in anesthetized cats, pointing towards an immediate effect of SMT on the activity of proprioceptive afferents. Proprioception is sub-served by mechanoreceptors on superficial and deep tissues. Located in the muscle belly parallel to the extrafusal muscle fibers, muscle spindles represent the main transmitters of proprioceptive information. Proprioceptive deficits have been suggested to provoke LBP through sensorimotor incongruence, abnormal loading across joint surfaces, and spinal instability due to less finely tuned muscular control, potentially causing sensorimotor dysfunction and degenerative processes in spinal tissues. In humans, there is anecdotal evidence that an SMT-induced repetitive barrage of proprioceptive input results in pain reduction and improves perceived function that might help to prevent LBP. However, a potential sustained and specific effect of SMT on lumbar proprioceptive function has not been systematically tested.

How one can test lumbar proprioceptive function in humans? Impairments in lumbar proprioception have been reported in LBP patients but only in sitting positions and mostly using proxy measures of proprioceptive function such as joint repositioning sense (JRS) and threshold to detect passive motion (TTDPM). The validity of these measures has been questioned as they measure position- and velocity-related proprioceptive sensation and the JRS is additionally influenced by motor skills and memory effects. Proprioceptive function can also be tested by assessing balance control (postural sway). Balance control presupposes a complex interplay involving the precise integration of proprioceptive inputs and motor outputs that can be tracked by analyzing postural sway on a force plate, a methodology that has been often used to assess differences in balance control in many diseases and conditions, including LBP. However, postural sway has been shown to be insensitive to changes of lumbar proprioceptive function, perhaps because postural sway relies on afferent input from various body locations and tissues. This can be overcome with a more direct assessment of proprioceptive function, achieved by using vibrotactile stimulation in combination with balance control measures. Vibration applied at frequencies between 60-80Hz (and amplitudes between 0.5-1mm) to muscles can selectively disturb proprioceptive signaling (mediated through primary (Ia) and secondary (II) muscle spindle afferents), affecting balance control by provoking corrective movements, often assessed through changes of the center of pressure (COP) in anterior-posterior direction. When endogenous or environmental conditions change, as in the instance of vibrotactile stimulation applied to the muscle, the balance control system must identify and selectively focus on sensory inputs providing the most reliable information, a process called sensory reweighting. Under normal conditions and while standing on a stable surface, healthy individuals rely on proprioceptive signals originating from ankle and paraspinal muscles. In contrast, standing on an unstable support surface (e.g. foam pad) forces individuals to rely less on ankle proprioception while up-weighting proprioceptive signals from paraspinal muscles. Differences in proprioceptive reweighting have been observed between healthy subjects and LBP patients by applying paraspinal and ankle muscle vibrotactile stimulation during a balance control task. Namely, during vibrotactile stimulation, individuals with recurrent LBP demonstrated an increased reliance on ankle proprioceptive signals compared to healthy subjects who up-weighted the proprioceptive signals from the paraspinal muscles (while down-weighting those from the ankle muscle to control postural balance). Importantly, a more "ankle-focused" strategy while standing on a stable support surface seems to increase the risk for developing or having recurrences of mild LBP within a time period of two years in young healthy individuals.

To test potential specific and sustained effects of SMT on lumbar proprioceptive function, the investigators aim to 1) assess SMT-induced changes in proprioceptive weighting (PW) over a two-week period and 2) use a rigorously controlled approach to control for non-specific effects. The planned experiments will be performed in healthy subjects and chronic LBP patients. This will allow to draw conclusions w.r.t. an isolated effect of SMT on lumbar proprioceptive function, providing a clear mechanism for SMT-induced changes in sensorimotor function.

ELIGIBILITY:
Inclusion criteria chronic LBP patients:

* Aged between 18 and 50
* History of chronic (>3months) LBP clinically not attributable to "red flags" (i.e., infection, trauma, fractures, inflammatory spondylarthropathies).
* Source of LBP clinically at the L4/5 or L5/S1 segment
* No history of vestibular disorders
* Body mass index (BMI) > 16 kg/m2

The presence of any one of the following exclusion criteria will lead to exclusion of the participant:

Exclusion criteria chronic LBP patients:

* Excessive consumption of alcohol or consumption of other drugs or analgesics within the last 24 h
* Pregnancy or breastfeeding
* Prior foot/ankle or spine surgery
* chiropractic (or other manual) treatment in the last 2 weeks
* facet joint, epidural or periradicular injections in the last 6 months
* any contraindication to spinal manipulative interventions (or are deemed unable to tolerate SMT to both body sides)
* Any neuromuscular diseases that might affect gait and posture and injuries of the motor system with permanent deformities
* Body mass index (BMI) > 30 kg/m2

Inclusion criteria healthy controls:

* Aged between 18 and 50
* No episode of musculoskeletal pain in the past 3 months
* No history of chronic pain (longer than 3 months)
* No history of vestibular disorders
* Body mass index (BMI) > 16 kg/m2

The presence of any one of the following exclusion criteria will lead to exclusion of the participant:

Exclusion criteria healthy controls:

* Excessive consumption of alcohol or consumption of other drugs or analgesics within the last 24 h
* Pregnancy or breastfeeding
* Prior foot/ankle or spine surgery
* chiropractic (or other manual) treatment in the last 2 weeks
* Any neuromuscular diseases that might affect gait and posture and injuries of the motor system with permanent deformities Body mass index (BMI) > 30 kg/m2

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 254 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Postural sway (mm) | 15 minutes
  Postural sway will be measured using a force plate system
Proprioceptive weighting ratio (value between 0 and 1) | 15 minutes
  The proprioceptive weighting ration will be calculated based on postural sway during vibrotactile stimulation on the ankle and paraspinal muscles

SECONDARY OUTCOMES:
Tampa-Scale for Kinesiophobia for the general population (TSK-G) questionnaire score | 10 minutes
  The original 17-item version of the TSK-G creates scores ranging between 17 and 68 higher scores indicating more fear of movement
Belief score influence of manipulation on balance control | 1 minute
  Subjects will be asked to rate how much they belief a manual intervention will affect their balance control (0 = no influence, 10 = maximal influence)
PainDETECT questionnaire | 5 minutes
  painDETECT is a nine-item questionnaire that consists of seven sensory symptom items for pain that are graded from 0= never to 5= strongly, one temporal item on pain-course pattern graded -1 to +1, and one spatial item on pain radiation graded 0 for no radiation or +2 for radiating pain
Pain intensity on numeric rating scale (NRS pain, 0-10) | 5 seconds
  Subjects will be ask to rate their current pain intensity on a scale ranging from 0 (no pain) to 10 (worst pain imaginable)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Chiropractic Medicine, University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No